CLINICAL TRIAL: NCT01553058
Title: A Trial to Determine the Effect of Psoriasis Treatment on Cardiometabolic Disease
Brief Title: Vascular Inflammation in Psoriasis Trial (The VIP Trial)
Acronym: VIP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 814278
Record Dates: First submitted 2012-02-14; First posted 2012-03-13 (Estimated); Results first posted 2018-05-22 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-04

CONDITIONS: Psoriasis; Cardiovascular Disease
Keywords: Psoriasis; Cardiovascular Disease; FDG/PET-CT; NB-UVB Phototherapy; Vascular Inflammation; Lipid Biomarkers
MeSH Terms: conditions — Psoriasis; Cardiovascular Diseases | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Adalimumab (Humira) (Active Comparator): Injection of the active drug Humira.
  Interventions: Drug: Adalimumab (Humira)
- Placebo Injection (Placebo Comparator): Injection of placebo in place of active Humira injection.
  Interventions: Drug: Placebo Injection
- NB-UVB phototherapy (Active Comparator): NB-UVB Phototherapy 3 times per week, no other intervention.
  Interventions: Other: NB-UVB phototherapy

INTERVENTIONS:
Drug: Adalimumab (Humira) — Humira will be given at an initial dose of 80mg followed by 40 mg the second week, subsequent doses will be given at 40mg and follow FDA dosing schedule.
  Arms: Adalimumab (Humira)
Drug: Placebo Injection — Placebo injection will be given according to the same dose and schedule as the active comparator.
  Arms: Placebo Injection
Other: NB-UVB phototherapy — Phototherapy will be given 3 times per week according to the Fitzpatrick scale for skin types.
  Arms: NB-UVB phototherapy

SUMMARY:
The purpose of this study is to assess the effect of adalimumab (Humira), when compared to NB-UVB (narrow-band ultraviolet B) phototherapy or placebo (an inactive substance that may resemble an active substance but has no medical value) injection. The study will compare the effects of each on systemic inflammation and cardiovascular disease risk factors in subjects diagnosed with moderate to severe psoriasis.

This study will look for systemic vascular inflammation in subjects with a test called FDG-PET/CT (Fluorodeoxyglucose-positron emission tomography/computed tomography). The study will also look for cardio metabolic (heart disease and metabolic factors such as diabetes) identifiers in the blood. A blood sample will be taken that will look for these markers identifying high cholesterol, cholesterol efflux function (the ability of cholesterol to move in the body), metabolic factors, and inflammation.

This study will also assess the effect of adalimumab (Humira), when compared to NB-UVB phototherapy or placebo injection on psoriasis activity and severity. The study will also compare the safety of adalimumab (Humira) to NB-UVB phototherapy or placebo injection. This study will also evaluate subjects' reported outcomes through a questionnaire that will assess quality-of-life in subjects living with psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 years of age and older.
2. Clinical diagnosis of psoriasis for at least 6 months as determined by subject interview of his/her medical history and confirmation of diagnosis through physical examination by Investigator.
3. Stable plaque psoriasis for at least 2 months before Screening and at Baseline (Week 0) as determined by subject interview of his/her medical history.
4. Moderate to severe psoriasis defined by ≥ 10 percent Body Surface Area (BSA) involvement at the Baseline (Week 0) visit.
5. PASI (psoriasis assessment and severity index) score of ≥ 12 at the Baseline (Week 0) visit.
6. Subject is a candidate for systemic therapy or phototherapy and has active psoriasis despite prior treatment with topical agents.
7. Women are eligible to participate in the study if they meet one of the following criteria:

   1. Women of childbearing potential who are willing to undergo regular pregnancy testing and agree to use one method of contraception throughout the study are eligible to participate
   2. Women who are postmenopausal (for at least one year), sterile, or hysterectomized are eligible to participate
   3. Women who have undergone tubal ligation are eligible to participate
   4. Women who agree to be sexually abstinent, defined as total abstinence from sexual intercourse, as a form of contraception are eligible to participate in the study.
8. Subject is judged to be in good general health as determined by the Principal Investigator based upon the results of medical history, laboratory profile, physical examination, and 12-lead electrocardiogram (ECG) performed at screening.
9. Able and willing to give written informed consent and to comply with requirements of this study protocol.

Exclusion Criteria:

1. Previous adverse event following exposure to a TNF-alpha antagonist and/or UV phototherapy that led to discontinuation of either of these therapies and contraindicates future treatment.
2. Previous lack of response to a TNF-alpha antagonist and/or UV phototherapy that led to discontinuation of either of these therapies.
3. Diagnosis of erythrodermic psoriasis, generalized or localized pustular psoriasis, medication-induced or medication-exacerbated psoriasis, or new onset guttate psoriasis.
4. Diagnosis of other active skin diseases or skin infections (bacterial, fungal, or viral) that may interfere with evaluation of psoriasis.
5. Cannot avoid UVB phototherapy for at least 14 days prior to the Baseline (Week 0) visit.
6. Cannot avoid psoralen-UVA phototherapy for at least 30 days prior to the Baseline (Week 0) visit and during the study.
7. Cannot discontinue systemic therapies for the treatment of psoriasis, or systemic therapies known to improve psoriasis, during the study:

   * Systemic (investigational or marketed) therapies must be discontinued at least 30 days prior to the Baseline (Week 0) visit except for biologics.

     * All biologics, except ustekinumab, must be discontinued for at least 90 days prior to Baseline (Week 0).
     * The IL-12/IL-23 antagonist ustekinumab (half-life of 45.6 ± 80.2 days) must be discontinued for at least 180 days prior to Baseline (Week 0).
   * Investigational agents must be discontinued at least 30 days or 5 half-lives (whichever is longer) prior to the Baseline (Week 0) visit.
8. Subject is taking or requires oral or injectable corticosteroids during the study. Inhaled corticosteroids for stable medical conditions are allowed.
9. Poorly controlled medical condition, such as unstable ischemic heart disease, congestive heart failure, recent cerebrovascular accidents, psychiatric disease requiring frequent hospitalization, and any other condition, which, in the opinion of the Investigator, would put the subject at risk by participation in the study.
10. History of diabetes mellitus, type 1 or type 2 - note that patients with type 2 diabetes may be enrolled if the duration of diabetes is <10 years and HbA1c is <7.0%)
11. Uncontrolled hypertension, with measured systolic blood pressure >180 mmHg or diastolic blood pressure >90 mmHg
12. History of demyelinating diseases or lupus.
13. Subject has infection or risk factors for severe infections, for example:

    * Positive serology or known history of HIV, hepatitis B or C, or other severe, recurrent, or persistent infections;
    * Excessive immunosuppression or other factors associated with it, including human immunodeficiency virus infection;
    * Active tuberculosis (TB) disease;
    * Evidence of latent TB infection demonstrated by Purified Protein Derivative (PPD) ≥ 5 mm of induration or positive Quantiferon-GOLD results; except if prophylactic treatment for TB, as recommended by local guidelines, is initiated prior to administration of study drug or if there is documentation that the subject has received prophylactic treatment for TB previously.
    * Any other significant infection requiring hospitalization or intravenous (IV) antibiotics in the month prior to Baseline;
    * Infection requiring treatment with oral or parenteral antibiotics within 14 days prior to Baseline;
    * Subject has received vaccination with Bacille Calmette-Guerin (BCG) within 365 days prior to Screening;
    * Subject has received vaccination with a live viral agent 30 days prior to Screening or will require a live vaccination during study participation including up to 30 days after the last dose of study drug.
14. Subject has history of hematological or solid malignancy other than successfully treated basal cell carcinoma, non-metastatic cutaneous squamous cell carcinoma or cervical carcinoma in situ.
15. Female subject who is pregnant or breast-feeding or considering becoming pregnant during the study.
16. Screening clinical laboratory analyses showing any of the following abnormal results:

    * Hemoglobin (Hgb) < 10 g/dL in females or <12 g/dL in males;
    * White blood cell (WBC) count <2.5 x 109/L

      o Subject can be included if WBC count is <2.5 x x 109/L and absolute neutrophil count (ANC) is >1000 cells / mm3.
    * WBC count > 15 x 109/L;
    * Platelet count < 100 x 109/L;
    * Serum aspartate transaminase (AST) or alanine transaminase (ALT) >2.5 upper limits of normal (ULN);
    * Serum total bilirubin ≥2 mg/dL (≥26 µmol/L); or
    * Serum creatinine >1.6 mg/dL (>141 µmol/L).
17. Recent history of substance abuse or psychiatric illness that could preclude compliance with the protocol.
18. History of any substance abuse within 365 days of screening visit
19. Alcohol use >14 drinks per week at the screening visit or within 30 days of the screening period
20. If subject is on cholesterol-lowering medication (e.g. statin), dose and form of medication must be stable for 90 days prior to week 0 and remain stable throughout the duration of the study.
21. History of photosensitivity of medical condition that may be exacerbated by UV exposures such as lupus or dermatomyositis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2012-07; Primary Completion 2016-08-08 (Actual); Study Completion 2016-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Gelfand, MD MSCE, Principal Investigator — University of Pennsylvania
Locations (9):
- United States (9):
  - University of California, Davis Health System, Sacramento, California
  - The University of Colorado, Denver, Colorado
  - National Heart, Lung, and Blood Institute, Bethesda, Maryland
  - Buffalo Medical Group, Buffalo, New York
  - Oregon Health & Science University, Portland, Oregon
  - The University of Pennsylvania, Philadelphia, Pennsylvania
  - Menter Dermatology Research Institute, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Noe MH, Wan MT, Shin DB, Armstrong AW, Duffin KC, Chiesa Fuxench ZC, Kalb RE, Menter A, Simpson EL, Takeshita J, Tyring SK, Van Voorhees AS, Mehta NN, Gelfand JM. Patient-reported outcomes of adalimumab, phototherapy, and placebo in the Vascular Inflammation in Psoriasis Trial: A randomized controlled study. J Am Acad Dermatol. 2019 Oct;81(4):923-930. doi: 10.1016/j.jaad.2019.05.080. Epub 2019 Jun 1. PMID 31163241
- [Derived] Mehta NN, Shin DB, Joshi AA, Dey AK, Armstrong AW, Duffin KC, Fuxench ZC, Harrington CL, Hubbard RA, Kalb RE, Menter A, Rader DJ, Reilly MP, Simpson EL, Takeshita J, Torigian DA, Werner TJ, Troxel AB, Tyring SK, Vanderbeek SB, Van Voorhees AS, Playford MP, Ahlman MA, Alavi A, Gelfand JM. Effect of 2 Psoriasis Treatments on Vascular Inflammation and Novel Inflammatory Cardiovascular Biomarkers: A Randomized Placebo-Controlled Trial. Circ Cardiovasc Imaging. 2018 Jun;11(6):e007394. doi: 10.1161/CIRCIMAGING.117.007394. PMID 29776990

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adalimumab (Humira) | Placebo Injection | NB-UVB Phototherapy
Started | 33 | 31 | 33
Completed | 32 | 30 | 30
Not Completed | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adalimumab (Humira) | Placebo Injection | NB-UVB Phototherapy | Total
Number analyzed (Participants) | 33 | 31 | 33 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.15 (13.97) | 44.32 (14.50) | 41.97 (13.97) | 43.46 (14.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 10 | 30
  Male | 24 | 20 | 23 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 7 | 15
  Not Hispanic or Latino | 27 | 28 | 26 | 81
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 2 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 3 | 9
  White | 27 | 24 | 26 | 77
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 2 | 5
Psoriasis Duration [Mean (Standard Deviation); unit: years] | 14.94 (14.73) | 19.29 (13.59) | 15.87 (13.55) | 16.7 (13.94)
Psoriatic Arthritis [Count of Participants; unit: Participants] | 4 | 2 | 3 | 9
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.93 (7.42) | 31.95 (7.74) | 32.61 (8.66) | 31.83 (7.91)
History of Cardiovascular Disease [Count of Participants; unit: Participants] | 2 | 3 | 2 | 7
Diabetes [Count of Participants; unit: Participants] | 3 | 1 | 0 | 4
Hypertension [Count of Participants; unit: Participants] | 6 | 7 | 5 | 18
Hyperlipidemia [Count of Participants; unit: Participants] | 5 | 5 | 4 | 14
Statin Use [Count of Participants; unit: Participants] | 1 | 4 | 3 | 8
10year Framingham Risk % [Mean (Standard Deviation); unit: percentage] — Absolute risk of developing a first cardiovascular disease (CVD) event (coronary death, myocardial infarction, coronary insufficiency, angina, ischemic stroke, hemorrhagic stroke, transient ischemic attack, peripheral artery disease, heart failure) within 10 years. The units are in 10-year risk percentage.
  percentage | 8.43 (7.75) | 7.91 (8.83) | 6.12 (7.68) | 7.53 (8.09)
Body Surface Area [Mean (Standard Deviation); unit: percentage] — Body Surface Area (BSA) is defined by how much (percentage) of the total body surface area is affected:
  Mild psoriasis: <5% of BSA Moderate psoriasis: 5-10% of BSA Severe psoriasis: >10% of BSA (Note: 1% of BSA is approximately equal to the palm of the patient's hand, excluding fingers)
  percentage | 23.39 (14.48) | 25.70 (15.02) | 22.96 (13.37) | 23.98 (14.19)
PASI (Psoriasis Area and Severity Index) [Mean (Standard Deviation); unit: units on a scale] — PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease).
  units on a scale | 18.89 (5.59) | 18.33 (7.64) | 19.32 (8) | 18.85 (7.08)
PGA (Physician's Global Assessment) [Mean (Standard Deviation); unit: units on a scale] — The PGA is an average assessment of all psoriatic lesions based on erythema, scale, and induration with score ranging from 0 (no evidence of disease) to 5 (maximal disease).
  units on a scale | 3.36 (.56) | 3.22 (.59) | 3.27 (.66) | 3.28 (.6)
DLQI (Dermatology Quality of Life Index) [Mean (Standard Deviation); unit: units on a scale] — The DLQI is calculated by summing the score of 10 questions regarding impact of skin condition on daily life resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
  units on a scale | 15.88 (5.53) | 13.48 (7.58) | 14.61 (6.52) | 14.68 (6.58)
History of Phototherapy [Count of Participants; unit: Participants] | 5 | 11 | 13 | 29
H/O Oral Systemics [Count of Participants; unit: Participants] | 10 | 10 | 11 | 31
H/O Biologics [Count of Participants; unit: Participants] | 10 | 11 | 8 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change in Vascular Inflammation
Description: Change in total vascular inflammation of five aortic segments as assessed on FDG-PET/CT between baseline and week 12. The arterial uptake of FDG is measured by the standardized uptake value (SUV) max divided by the venous SUV mean yielding a target to background ratio (TBR).
Time Frame: Baseline - Week 12
Measure: Mean (Standard Deviation); unit: Tissue-to-background ratio (TBR)
Arm/Group | Adalimumab (Humira) | Placebo Injection | NB-UVB Phototherapy
Number analyzed (Participants) | 33 | 31 | 33
Tissue-to-background ratio (TBR) | -.067 (.213) | -.052 (.112) | -.079 (.020)
Statistical Analysis 1: Comparison: Adalimumab (Humira) vs Placebo Injection; Test type: Other — Difference of Differences; p = 0.795, Regression, Linear
Statistical Analysis 2: Comparison: Placebo Injection vs NB-UVB Phototherapy; Test type: Other — Difference of differences; p = 0.647, Regression, Linear

2. Primary Outcome: Change in Cardiometabolic Biomarkers: Total Cholesterol
Description: To assess the effects of adalimumab, as compared to NB-UVB phototherapy or placebo, in patients with moderate to severe psoriasis on total cholesterol.
Time Frame: Baseline - Week 12
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Adalimumab (Humira): Injection of the active drug Humira. Adalimumab (Humira): Humira will be given at an initial dose of 80mg followed by 40 mg the second week, subsequent doses will be given at 40mg and follow FDA dosing schedule.
- Placebo Injection: Injection of placebo in place of active Humira injection. Placebo Injection: Placebo injection will be given according to the same dose and schedule as the active comparator.
- NB-UVB Phototherapy: NB-UVB Phototherapy 3 times per week, no other intervention. NB-UVB phototherapy: Phototherapy will be given 3 times per week according to the Fitzpatrick scale for skin types.
Arm/Group | Adalimumab (Humira) | Placebo Injection | NB-UVB Phototherapy
Number analyzed (Participants) | 33 | 31 | 33
mg/dL | 1.48 (21.25) | 5.00 (25.22) | 3.15 (32.81)
Statistical Analysis 1: Comparison: Adalimumab (Humira) vs Placebo Injection; Test type: Other — Difference of differences; p = 0.386, Regression, Linear
Statistical Analysis 2: Comparison: Placebo Injection vs NB-UVB Phototherapy; Test type: Other — Difference of Differences; p = 0.280, Regression, Linear

3. Secondary Outcome: Change in Psoriasis Activity (PASI-75 and PGA)
Description: Psoriasis activity will be assessed using standard psoriasis measurements, PASI75 and PGA Clear/Almost Clear
Time Frame: Baseline - Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab (Humira) | Placebo Injection | NB-UVB Phototherapy
Number analyzed (Participants) | 32 | 30 | 30
Participants
  PASI75 | 15 | 2 | 14
  PGA Clear/Almost Clear | 14 | 2 | 8

4. Secondary Outcome: Change in Patient-reported Outcomes-EuroQol EQ-5D
Description: EQ-5D is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. The EQ-5D consists of a descriptive system and the EQ VAS. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression on a scale ranging from 1 (no health state problem) to 3 (extreme health state problems). The EQ VAS records the patient's self-rated health on a vertical visual analogue scale ranging from 0, worst health state, to 100, best health state. A scoring function is used to assign a value (i.e., EQ-5D™ index score) to self-reported health states from a set of population-based preference weights. For the U.S. general population, the possible EQ-5D index scores range from -0.11 to 1.0 where 0.0 = death and 1.0 = perfect health.
Time Frame: Baseline -Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab (Humira) | Placebo Injection | NB-UVB Phototherapy
Number analyzed (Participants) | 33 | 31 | 33
units on a scale | .07 (.14) | .0 (.17) | .16 (.19)

5. Secondary Outcome: Change in Patient-reported Outcomes-Dermatology Life Quality Index (DLQI)
Description: Patient reported quality of life outcomes will be assessed using DLQI. The DLQI is calculated by summing the score of 10 questions regarding impact of skin condition on daily life resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Time Frame: Baseline - Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab (Humira) | Placebo Injection | NB-UVB Phototherapy
Number analyzed (Participants) | 33 | 31 | 33
units on a scale | -7.91 (8.77) | -3.73 (8) | -9.27 (4.70)

6. Secondary Outcome: Change in Patient-reported Outcomes-MEDFICTS Dietary Assessment)
Description: Patient reported dietary outcomes will be assessed using MEDFICTS (Meats, Eggs, Dairy, Fried foods, fat In baked goods, Convenience foods, fats added at the Table, and Snacks), a brief dietary assessment instrument for properly assessing cardiovascular diet. The questionnaire yields a continuous score (ranging from 0 to 216), with a score of <40 indicating adherence to the Therapeutic Lifestyle Changes (TLC) diet (intake of <7% of energy from saturated fat, <30% of energy from total fat, and <200 mg dietary cholesterol/day).
Time Frame: Baseline to Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab (Humira) | Placebo Injection | NB-UVB Phototherapy
Number analyzed (Participants) | 33 | 31 | 33
units on a scale | -10.17 (17.47) | -13.66 (28.59) | -16.29 (20.94)

7. Secondary Outcome: Change in Patient-reported Outcomes-International Physical Activity Questionnaire (IPAQ)
Description: Patient reported physical activity will be assessed using IPAQ. IPAQ is an instrument designed primarily for population surveillance of physical activity among adults with activity measured in metabolic equivalent (MET)-minutes per week.
Time Frame: Baseline week 4, 8 and 12
Measure: Mean (Standard Deviation); unit: MET-minutes/week
Arm/Group | Adalimumab (Humira) | Placebo Injection | NB-UVB Phototherapy
Number analyzed (Participants) | 33 | 31 | 33
MET-minutes/week | 1282 (4837) | 141 (2921) | 18 (2994)

8. Secondary Outcome: Number of Patients With Adverse Events.
Description: Safety will be assessed by comparing how many patients have adverse events depending on whether they are on adalimumab, as compared to NB-UVB phototherapy or placebo.
Time Frame: Baseline - Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab (Humira) | Placebo Injection | NB-UVB Phototherapy
Number analyzed (Participants) | 33 | 31 | 33
Participants
  erythema | 0 | 0 | 14
  pruritis | 0 | 0 | 6
  photosensitivity | 0 | 0 | 3
  upper respiratory infection | 3 | 4 | 2
  nasal congestion | 1 | 1 | 2
  cough | 0 | 2 | 0
  sore throat | 0 | 2 | 1
  headache | 1 | 2 | 2
  myalgia | 0 | 2 | 1
  joint range of motion decrease | 2 | 0 | 0
  depression | 0 | 0 | 2
  tooth infection | 0 | 2 | 0

9. Primary Outcome: Change in Cardiometabolic Biomarkers: Cholesterol Efflux
Description: To assess the effects of adalimumab, as compared to NB-UVB phototherapy or placebo, in patients with moderate to severe psoriasis on cholesterol efflux capacity. The ability to promote cholesterol efflux from macrophages is a classic function of HDL that is thought to be an important mechanism by which HDL protects against atherosclerosis. HDL cholesterol efflux capacity assays are performed based on published methods using J774 cells derived from a murine macrophage cell line (Mehta NN Atherosclerosis 2012). Efflux is calculated as a unitless measure by using the following formula: [(µCi of 3H-cholesterol in media containing apoB-depleted subject plasma - µCi of 3H-cholesterol in plasma-free media) / (µCi of 3H-cholesterol in media containing apoB-depleted pooled control plasma-µCi of 3H-cholesterol in pooled control plasma-free media)]. The pooled plasma was obtained from five healthy volunteers.
Time Frame: Baseline - Week 12
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Adalimumab (Humira) | Placebo Injection | NB-UVB Phototherapy
Number analyzed (Participants) | 33 | 31 | 33
unitless | 0.05 (0.25) | 0.00 (0.15) | 0.04 (0.16)
Statistical Analysis 1: Comparison: Adalimumab (Humira) vs Placebo Injection; Test type: Other — Difference of Differences; p = 0.357, Regression, Linear
Statistical Analysis 2: Comparison: Placebo Injection vs NB-UVB Phototherapy; Test type: Other — Difference of Differences; p = 0.496, Regression, Linear

10. Primary Outcome: Change in Cardiometabolic Biomarkers: Low Density Lipoprotein Particle Total
Description: To assess the effects of adalimumab, as compared to NB-UVB phototherapy or placebo, in patients with moderate to severe psoriasis on low density lipoprotein particle total.
Time Frame: Baseline - Week 12
Measure: Mean (Standard Deviation); unit: nmol/L
Groups:
- Placebo Injection: njection of placebo in place of active Humira injection. Placebo Injection: Placebo injection will be given according to the same dose and schedule as the active comparator.
Arm/Group | Adalimumab (Humira) | Placebo Injection | NB-UVB Phototherapy
Number analyzed (Participants) | 33 | 31 | 33
nmol/L | -25.70 (263.32) | -34.90 (319.42) | 17.42 (187.63)
Statistical Analysis 1: Comparison: Adalimumab (Humira) vs Placebo Injection; Test type: Other — Difference of Differences; p = 0.897, Regression, Linear
Statistical Analysis 2: Comparison: Placebo Injection vs NB-UVB Phototherapy; Test type: Other — Difference of differences; p = 0.467, Regression, Linear

11. Primary Outcome: Change in Cardiometabolic Biomarkers: High Density Lipoprotein Particle Total
Description: To assess the effects of adalimumab, as compared to NB-UVB phototherapy or placebo, in patients with moderate to severe psoriasis on high density lipoprotein particle total.
Time Frame: Baseline - Week 12
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Adalimumab (Humira) | Placebo Injection | NB-UVB Phototherapy
Number analyzed (Participants) | 33 | 31 | 33
umol/L | 0.59 (4.00) | -1.97 (7.03) | 1.35 (5.06)
Statistical Analysis 1: Comparison: Adalimumab (Humira) vs Placebo Injection; Test type: Other — Difference of differences; p = 0.089, Regression, Linear
Statistical Analysis 2: Comparison: Placebo Injection vs NB-UVB Phototherapy; Test type: Other — Difference of differences; p = 0.030, Regression, Linear

12. Primary Outcome: Change in Cardiometabolic Biomarkers: Log Insulin
Description: To assess the effects of adalimumab, as compared to NB-UVB phototherapy or placebo, in patients with moderate to severe psoriasis on log insulin.
Time Frame: Baseline - Week 12
Measure: Mean (Standard Deviation); unit: log(pg/mL)
Arm/Group | Adalimumab (Humira) | Placebo Injection | NB-UVB Phototherapy
Number analyzed (Participants) | 33 | 31 | 33
log(pg/mL) | -0.19 (0.71) | -0.21 (0.74) | -0.13 (0.46)
Statistical Analysis 1: Comparison: Adalimumab (Humira) vs Placebo Injection; Test type: Other — Difference of differences; p = 0.934, Regression, Linear
Statistical Analysis 2: Comparison: Placebo Injection vs NB-UVB Phototherapy; Test type: Other — Difference of differences; p = 0.679, Regression, Linear

13. Primary Outcome: Change in Cardiometabolic Biomarkers: Log Adiponectin
Description: To assess the effects of adalimumab, as compared to NB-UVB phototherapy or placebo, in patients with moderate to severe psoriasis on log adiponectin.
Time Frame: Baseline - Week 12
Measure: Mean (Standard Deviation); unit: log(ug/mL)
Arm/Group | Adalimumab (Humira) | Placebo Injection | NB-UVB Phototherapy
Number analyzed (Participants) | 33 | 31 | 33
log(ug/mL) | -0.07 (2.05) | 0.07 (0.45) | -0.08 (.41)
Statistical Analysis 1: Comparison: Adalimumab (Humira) vs Placebo Injection; Test type: Other — Difference of differences; p = 0.672, Regression, Linear
Statistical Analysis 2: Comparison: Placebo Injection vs NB-UVB Phototherapy; Test type: Other — Difference of differences; p = 0.655, Regression, Linear

14. Primary Outcome: Change in Cardiometabolic Biomarkers: Log Leptin
Description: To assess the effects of adalimumab, as compared to NB-UVB phototherapy or placebo, in patients with moderate to severe psoriasis on log leptin.
Time Frame: Baseline - Week 12
Measure: Mean (Standard Deviation); unit: log(pg/mL)
Arm/Group | Adalimumab (Humira) | Placebo Injection | NB-UVB Phototherapy
Number analyzed (Participants) | 33 | 31 | 33
log(pg/mL) | -0.06 (0.55) | 0.03 (0.47) | 0.08 (0.42)
Statistical Analysis 1: Comparison: Adalimumab (Humira) vs Placebo Injection; Test type: Other — Difference of differences; p = 0.504, Regression, Linear
Statistical Analysis 2: Comparison: Placebo Injection vs NB-UVB Phototherapy; Test type: Other — Difference of differences; p = 0.695, Regression, Linear

15. Primary Outcome: Change in Cardiometabolic Biomarkers: Log C-reactive Protein
Description: To assess the effects of adalimumab, as compared to NB-UVB phototherapy or placebo, in patients with moderate to severe psoriasis on log C-reactive protein (CRP).
Time Frame: Baseline - Week 12
Measure: Mean (Standard Deviation); unit: log(pg/mL)
Arm/Group | Adalimumab (Humira) | Placebo Injection | NB-UVB Phototherapy
Number analyzed (Participants) | 33 | 31 | 33
log(pg/mL) | -0.52 (1.00) | 0.35 (1.06) | -0.50 (1.14)
Statistical Analysis 1: Comparison: Adalimumab (Humira) vs Placebo Injection; Test type: Other — Difference of differences; p = 0.002, Regression, Linear
Statistical Analysis 2: Comparison: Placebo Injection vs NB-UVB Phototherapy; Test type: Other — Difference of differences; p = 0.009, Regression, Linear

16. Primary Outcome: Change in Cardiometabolic Biomarkers: Log Tumor Necrosis Factor-alpha
Description: To assess the effects of adalimumab, as compared to NB-UVB phototherapy or placebo, in patients with moderate to severe psoriasis on log Tumor necrosis factor-alpha.
Time Frame: Baseline - Week 12
Measure: Mean (Standard Deviation); unit: log(pg/mL)
Arm/Group | Adalimumab (Humira) | Placebo Injection | NB-UVB Phototherapy
Number analyzed (Participants) | 33 | 31 | 33
log(pg/mL) | -0.27 (0.33) | 0.14 (0.38) | -0.04 (0.36)
Statistical Analysis 1: Comparison: Adalimumab (Humira) vs Placebo Injection; Test type: Other — Difference of Differences; p < 0.001, Regression, Linear
Statistical Analysis 2: Comparison: Placebo Injection vs NB-UVB Phototherapy; Test type: Other — Difference of differences; p = 0.065, Regression, Linear

17. Primary Outcome: Change in Cardiometabolic Biomarkers: Log Interleukin 6
Description: To assess the effects of adalimumab, as compared to NB-UVB phototherapy or placebo, in patients with moderate to severe psoriasis on log interleukin 6.
Time Frame: Baseline - Week 12
Measure: Mean (Standard Deviation); unit: log(pg/mL)
Arm/Group | Adalimumab (Humira) | Placebo Injection | NB-UVB Phototherapy
Number analyzed (Participants) | 33 | 31 | 33
log(pg/mL) | -0.57 (1.08) | 0.20 (0.99) | -0.49 (1.08)
Statistical Analysis 1: Comparison: Adalimumab (Humira) vs Placebo Injection; Test type: Other — Difference of differences; p = 0.007, Regression, Linear
Statistical Analysis 2: Comparison: Placebo Injection vs NB-UVB Phototherapy; Test type: Other — Difference of differences; p = 0.019, Regression, Linear

18. Primary Outcome: Change in Cardiometabolic Biomarkers: GlycA
Description: To assess the effects of adalimumab, as compared to NB-UVB phototherapy or placebo, in patients with moderate to severe psoriasis on GlycA
Time Frame: Baseline - Week 12
Measure: Mean (Standard Deviation); unit: log(pg/mL)
Arm/Group | Adalimumab (Humira) | Placebo Injection | NB-UVB Phototherapy
Number analyzed (Participants) | 33 | 31 | 33
log(pg/mL) | -35.89 (40.38) | 5.28 (66.83) | -1.92 (52.89)
Statistical Analysis 1: Comparison: Adalimumab (Humira) vs Placebo Injection; Test type: Other — Difference of differences; p = 0.006, Regression, Linear
Statistical Analysis 2: Comparison: Placebo Injection vs NB-UVB Phototherapy; Test type: Other — Difference of differences; p = 0.628, Regression, Linear

ADVERSE EVENTS:
Time Frame: Baseline - Week 12
Arm/Group | Adalimumab (Humira) | Placebo Injection | NB-UVB Phototherapy
Serious Adverse Events (participants affected / at risk) | 2/33 | 0/31 | 0/33
Other Adverse Events (participants affected / at risk) | 7/33 | 15/31 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab (Humira) (N=33) | Placebo Injection (N=31) | NB-UVB Phototherapy (N=33)
vasovagal syncope (General disorders) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab (Humira) (N=33) | Placebo Injection (N=31) | NB-UVB Phototherapy (N=33)
pruritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 6 (6)
erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 14 (14)
photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
upper respiratory infection (Infections and infestations) | 3 (3) | 4 (4) | 2 (2)
nasal congestion (General disorders) | 1 (1) | 1 (1) | 2 (2)
cough (General disorders) | 0 (0) | 2 (2) | 0 (0)
sore throat (General disorders) | 0 (0) | 2 (2) | 1 (1)
headache (General disorders) | 1 (1) | 2 (2) | 2 (2)
myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
joint range of motion decrease (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
tooth infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes